CLINICAL TRIAL: NCT01667861
Title: Risk Factors for Glaucoma in Musicians
Status: Completed | Type: Observational
Sponsor: Henny Beckers (Other)
Collaborators: Stichting Glaucoomfonds (Unknown)
Responsible Party: Sponsor-Investigator, Henny Beckers, MD, PhD, FEBophth, Maastricht University Medical Center
Organization: Maastricht University Medical Center (Other)
Other Study IDs: NL25853.068.09/MEC09-2-112
Record Dates: First submitted 2012-08-10; First posted 2012-08-17 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Glaucoma
Keywords: Glaucoma; Wind instruments
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- (Wind) musicians: Members of (professional) orchestras, especially wind instrument players.

SUMMARY:
The purpose of this study is to determine the impact of playing wind instruments for the development of ocular hypertension and glaucoma, together with investigating the prevalence of visual problems and eye diseases in (professional) musicians.

ELIGIBILITY:
Inclusion Criteria:

* All full time or part time professional players of participating symphony or wind orchestras, including guest players.
* Retired players, if possible.

Exclusion Criteria:

* Difficulty in reading or speaking Dutch.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: (Professional) musicians, who play in symphony or wind orchestras.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
IOP levels, including IOP peaks occurring during or directly after playing, and prevalence of glaucomatous field loss in players of wind instruments. | One hour.
IOP peaks and variations during continuous IOP monitoring | 24 hours
  Several high-risk participants will be asked their permission to perform continuous IOP monitoring during 24 hours with a sensing contact lens.

SECONDARY OUTCOMES:
Risk factors for glaucoma and the prevalence of visual problems and eye disease among (professional) musicians | 2 years
  Participants of orchestras will be asked to fill in a questionnaire to collect demographic data together with data on musical history,ophthalmologic history and family history on glaucoma and ocular hypertension. From these participants, a selection will be invited for further screening.

CONTACTS AND LOCATIONS:
Overall Officials: Henny JM Beckers, MD, PhD, Principal Investigator — Maastricht University Medical Center, NL
Locations (1):
- University Eye Clinic, Maastricht University Medical Center, Maastricht, Netherlands